CLINICAL TRIAL: NCT02591095
Title: A Study of ABT-263 as Single Agent in Women With Platinum Resistant/Refractory Recurrent Ovarian Cancer
Acronym: MONAVI-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: ARCAGY/ GINECO GROUP (Other); French Cancer Research Hospital Program (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-000193-35
Record Dates: First submitted 2015-10-14; First posted 2015-10-29 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Platinum-resistant or Refractory Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — navitoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ABT-263 (Experimental): oral Navitoclax (ABT-263) daily
  Interventions: Drug: ABT-263

INTERVENTIONS:
Drug: ABT-263

SUMMARY:
ABT-263 as single agent in women with platinum resistant/refractory recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* - Woman older than 18 years
* Subjects with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Histologically and/or cytologically documented high grade serous epithelial cancer of ovarian, fallopian tube or peritoneum
* Platinum resistant ovarian cancer defined as relapsing within 6 months after a platinum based chemotherapy OR platinum refractory ovarian cancer defined as progressing during a platinum based chemotherapy (excepted refractory patients in first line)
* Subjects having received at least 2 prior lines of treatments including platinum regimen
* Subjects who are willing and able to comply with the protocol and study procedures including willingness to undergo tumor biopsy before therapy at screening
* There is no limitation to prior number of therapies
* Patients must have documented disease progression
* Subjects who have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Adequate bone marrow, renal and hepatic function per local laboratory reference range as follows:• Absolute Neutrophil Count ≥ 1500/ mm3

  * Platelets ≥ 150,000 / mm3
  * Hemoglobin ≥ 9.0 g/dL
  * Renal function: Serum creatinine ≤1.2mg/dL or calculated creatinine clearance ≥ 60mL/min
  * AST/ALT ≤ 3.0× the upper limit of normal (ULN); [Subjects with liver metastasis may have AST, ALP, and ALT less then or equal to 5.0 X ULN]
  * Bilirubin ≤ 1.25×ULN
  * Coagulation: aPTT and PT not to exceed 1.2 × ULN
* LVEF > 50% by echocardiograms or MUGA
* Patients must give written informed consent

Exclusion Criteria:

* Patient's refusal or impossibility to perform biopsy on relapsing disease
* Bowel occlusive syndrome or other gastro-intestinal disorder that does not allow oral medication such as malabsorption
* Patients with platinum refractory disease in first line
* Received radio-immunotherapy within 6 months of 1st dose of study drug
* Received steroid therapy for anti-neoplastic intent within 7 days of the 1st dose of study drug (Inhaled steroids for asthma, topical steroids, replacement/stress corticosteroids, or corticosteroids taken as premedication are allowed)
* Consumption of grapefruit or grapefruit products within 3 days prior to the first dose of study drug
* Patient receiving treatments strong CYP3A4 inhibitors or inducers (Appendix A)
* Positive for HIV and VHC
* Predisposing condition/currently exhibiting signs of bleeding
* Currently receiving anticoagulation therapy, exception of low-dose anticoagulation medications for prophylaxis
* Received aspirin within 7 days of start dose of study drug
* Active peptic ulcer disease / other potentially hemorrhagic esophagitis/gastritis
* Active immune thrombocytopenic purpura, autoimmune hemolytic anemia or history of being refractory to platelet transfusions (within 1 year of 1st dose of study drug)
* Uncontrolled cardiac, renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease, active systemic fungal infection; diagnosis of fever and neutropenia within 1 week of study drug administration
* A evidence of current/active malignancies other than ovarian cancer
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the progression-free survival (PFS) in the whole cohort of patients with a recurrent platinum-resistant ovarian cancer. | the time to progression (or death from any cause) from date of randomization until date of first documented progression or date of death from any cause,whichever came first, assessed up to 12 months. Evaluation at interim and final analyses.

SECONDARY OUTCOMES:
Bim expression level | biopsy sample before initiation of treatment by ABT-263 and assessment within 6 months after end of inclusions
  Bim expression level expressed by immunohistochemistry on biopsy of relapsing tumor at inclusion
Response rate | evaluated every 6 weeks during treatment to progression or death for any cause.(during average 12 months)]
  - Response rate defined by a complete response (CR), a partial response (PR) or a stable disease (SD) according to the RECIST v1.1
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months.
Incidence of Treatment-Emergent Adverse Events according to the NCI CTC AE version 4.0 | From date of treatment start until end of study participation (during average 12 months)]
  Toxicities
Peak Plasma Concentration of ABT-263 | 8-hour post-dose PK on D1 of C1 & 2. Dosage will be done within 12 months after end of inclusions
Residual concentration of ABT-263 | Pre-dose 0 and cycles 3, 4, 6 . Dosage will be done within 12 months after end of inclusions

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CHU, Lyon
  - ICM Val d'Aurelle, Montpellier
  - ICL Institut de Cancérologie de Lorraine, Nancy
  - Centre Catherine de Sienne, Nantes
  - ICO Centre René Gauducheau, Nantes
  - ICO Paul Papin, Nantes
  - Centre Antoine LACASSAGNE, Nice
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Joly F, Fabbro M, Follana P, Lequesne J, Medioni J, Lesoin A, Frenel JS, Abadie-Lacourtoisie S, Floquet A, Gladieff L, You B, Gavoille C, Kalbacher E, Briand M, Brachet PE, Giffard F, Weiswald LB, Just PA, Blanc-Fournier C, Leconte A, Clarisse B, Leary A, Poulain L. A phase II study of Navitoclax (ABT-263) as single agent in women heavily pretreated for recurrent epithelial ovarian cancer: The MONAVI - GINECO study. Gynecol Oncol. 2022 Apr;165(1):30-39. doi: 10.1016/j.ygyno.2022.01.021. Epub 2022 Feb 2. PMID 35123771